CLINICAL TRIAL: NCT00468715
Title: Bicalutamide for the Treatment of Androgen Receptor Positive (AR(+)), Estrogen Receptor Negative, Progesterone Receptor Negative (ER(-)/PR(-)) Metastatic Breast Cancer Patients: A Phase II Feasibility Study
Brief Title: Bicalutamide in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-022; MSKCC-07022
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — bicalutamide; Immunohistochemistry

ARMS (1):
- bicalutamide (Experimental): This is a multicenter, open-label, phase II study to evaluate the antitumor activity and safety of bicalutamide administered orally daily to patients with ER(-)/PR(-)/AR(+) metastatic breast cancer. Eligible patients who have consented to trial participation will receive bicalutamide at a dose of 150mg PO daily.
  Interventions: Drug: bicalutamide; Other: diagnostic laboratory biomarker analysis; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: bicalutamide
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Androgens can cause the growth of breast cancer cells. Antihormone therapy, such as bicalutamide, may stop the adrenal glands from making androgens.

PURPOSE: This phase II trial is studying how well bicalutamide works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 6-month efficacy rate of bicalutamide as first-, second-, or third-line therapy in patients with androgen receptor-positive and estrogen receptor- and progesterone receptor-negative metastatic breast cancer.

Secondary

* Determine the 6-month progression-free survival of patients treated with this drug.
* Evaluate the safety of this drug in these patients.
* Evaluate changes in estradiol, total and free testosterone, and sex-hormone binding globulin in response to androgen blockade in patients treated with this drug.
* Evaluate tissue, including cytokeratins 5/6 and 17, SPDEF, ALCAM, ERBB2, FGFR4, and prostate-specific antigen (PSA), using immunohistochemical analysis in patients treated with this drug.

OUTLINE: This is a open-label study.

Patients receive oral bicalutamide once daily for 4 weeks. Treatment repeats every 4 weeks for 6 months in the absence of disease progression or unacceptable toxicity. Patients achieving complete response, partial response, or stable disease may continue to receive bicalutamide as above at the discretion of the investigator.

Patients undergo blood and tissue sample collection for correlative studies. Samples are analyzed for hormonal levels, including estradiol, total testosterone, free testosterone, and sex-hormone binding globulin, and proteins, including ALCAM, SPEDF, and CK 5/6, by immunohistochemical analysis at baseline, after course 1, and at the end of the study.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Stage IV disease
* Measurable or non-measurable disease
* Patients with HER2/neu-positive disease must have received prior trastuzumab (Herceptin®)
* No active brain metastases or leptomeningeal disease

  * History of brain metastases allowed provided lesions are stable for at least 3 months as documented by head CT scan or MRI of the brain
* Hormone receptor status:

  * Estrogen receptor- and progesterone receptor-negative*
  * Androgen receptor-positive* NOTE: *Samples are considered positive if greater than 10% of cell nuclei are immunoreactive

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (unless bone metastases are present in the absence of liver metastases)
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious medical or psychiatric illness
* No serious active infection
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No hypersensitivity reaction to bicalutamide or any of the tablet's components

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior cytotoxic chemotherapy and recovered
* At least 3 weeks since prior investigational drugs
* At least 4 weeks since prior major surgery and recovered
* Prior neoadjuvant or adjuvant chemotherapy allowed

  * Any number of chemotherapy regimens are allowed for metastatic disease
* Prior hormonal therapy allowed
* No concurrent chemotherapy, other hormonal therapy, immunotherapy, or biological therapy
* No concurrent trastuzumab (Herceptin®)
* No concurrent enrollment in another clinical trial in which investigational procedures are performed or investigational therapies are administered

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-03-23 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany A. Traina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bicalutamide: This is a multicenter, open-label, phase II study to evaluate the antitumor activity and safety of bicalutamide administered orally daily to patients with ER(-)/PR(-)/AR(+) metastatic breast cancer. Eligible patients who have consented to trial participation will receive bicalutamide at a dose of 150mg PO daily.
  bicalutamide
  diagnostic laboratory biomarker analysis
  immunohistochemistry staining method
Period: Overall Study
Arm/Group | Bicalutamide
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bicalutamide
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 54 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: 6-month Response Rate (Complete Response, Partial Response, and Stable Disease)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bicalutamide
Number analyzed (Participants) | 28
Participants
  Stable Disease | 9
  Progression of Disease | 15
  Not Entered | 4

2. Secondary Outcome: Count of Participants With Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bicalutamide
Number analyzed (Participants) | 28
Participants
  Participants who progressed | 22
  Participants who did not progress | 6

3. Secondary Outcome: Number of Participants Evaluated for Toxicity
Description: Toxicity measured by CTCAE v3.0
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bicalutamide
Number analyzed (Participants) | 28
Participants | 28

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bicalutamide
All-Cause Mortality (participants affected / at risk) | 14/28
Serious Adverse Events (participants affected / at risk) | 4/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bicalutamide (N=28)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Blood/Bone Marrow, other (Blood and lymphatic system disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Colitis, infection (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 1
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 4
Lymphopenia (Investigations) | 1
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 4
Mood alteration - Depression (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pain - abdomen NOS (Gastrointestinal disorders) | 1
Pain - back (Musculoskeletal and connective tissue disorders) | 1
Phospate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 4
Platelets (Investigations) | 1
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bicalutamide (N=28)
AST, SGOT (Investigations) | 10
Fatigue (General disorders) | 9
ALT, SGPT (Investigations) | 8
Edema, limb (General disorders) | 8
Hot flashes/flushes (Vascular disorders) | 7
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 6
Hemoglobin (Blood and lymphatic system disorders) | 6
Alkaline Phosphatase (Investigations) | 5
Constipation (Gastrointestinal disorders) | 5
Leukocytes (total WBC) (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Bilirubin (hyperbilirubinemia) (Investigations) | 4
Nausea (Gastrointestinal disorders) | 4
Neuropathy, sensory (Nervous system disorders) | 4
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 3
Pain - breast (Reproductive system and breast disorders) | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Platelets (Investigations) | 3
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Investigations) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 2
Mood alteration - Anxiety (Psychiatric disorders) | 2
Mood alteration - Depression (Psychiatric disorders) | 2
Ocular/visual - other (Eye disorders) | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Bone (Musculoskeletal and connective tissue disorders) | 2
Pain - other (specify) (General disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT00468715/Prot_SAP_000.pdf